CLINICAL TRIAL: NCT05442463
Title: Hormone Therapy and Angiotensin-Dependent Arterial and Renal
Brief Title: Hormone Therapy and Angiotensin-Dependent Arterial and Renal Vasoconstriction in Humans
Status: Recruiting | Type: Observational
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Sofia Ahmed, Principal Investigator, University of Calgary
Other Study IDs: REB19-0460
Record Dates: First submitted 2022-06-28; First posted 2022-07-05 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Hormone Therapy
Keywords: post menopausal hormone replacement therapy; transgender men; transgender women; nonbinary; cis gender; post menopause; HRT; hormone replacement therapy
MeSH Terms: interventions — Captopril; Iohexol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine, blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cisgender and transgender women: Iohexol 5 ml IV push followed 10 ml IV flush of normal saline is administered to establish baseline GFR (glomerular filtration rate). FF (filtration fraction) is calculated as follows: GFR/RPF=FF. Captopril 25 mg is given orally.
  Blood will be collected at specific time points, pulse wave velocity testing 3 times throughout morning, Holter monitor and bioelectrical impedance testing.
  Interventions: Drug: Captopril Tablets; Drug: Iohexol
- Cisgender and transgender men: Iohexol 5 ml IV push followed 10 ml IV flush of normal saline is administered to establish baseline GFR (glomerular filtration rate). FF (filtration fraction) is calculated as follows: GFR/RPF=FF. Captopril 25 mg is given orally.
  Blood will be collected at specific time points, pulse wave velocity testing 3 times throughout morning, Holter monitor and bioelectrical impedance testing.
  Interventions: Drug: Captopril Tablets; Drug: Iohexol

INTERVENTIONS:
Drug: Captopril Tablets — Captorpril challenge to each participant
  Other Names: Capoten
Drug: Iohexol — Iohexol infusion to evaluate measured GFR
  Other Names: Omnipaque

SUMMARY:
1. to investigate the association between route of administration of exogenous estrogen (transdermal vs. oral) and cardiorenal risk in cisgender (gender identity aligning with sex at birth) and transgender (gender identity not aligning with sex at birth) women.
2. to investigate the association between exogenous testosterone exposure and cardiorenal risk in cisgender (gender identity aligning with sex at birth) and transgender (gender identity not aligning with sex at birth) men.

DETAILED DESCRIPTION:
Participants are screened for eligibility.

Study involves a 4.5 hour morning in the lab:

1. Participants come fasting
2. IV infusion and blood draws
3. Non invasive testing - Holter monitor, sphygmocor, bioelectrical impedance, blood pressure checks

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 90 years
* Taking hormones orally or non-orally (either estrogen, progesterone or testosterone)

Exclusion Criteria:

* Cardiovascular disease (symptoms consistent with myocardial ischemia, previously documented myocardial ischemia, cardiac arrhythmias or valve abnormalities, or abnormal ECG at screening)
* Cerebrovascular disease (transient ischemic attacks or stroke)
* History of hypertension (BP>140/90 or use of antihypertensive medications)
* Estimated glomerular filtration rate (eGFR) < 60 ml/min/1.73m2
* Diabetes mellitus (defined by history, use of hypoglycaemic agents or a fasting glucose >7mmol/L)
* Current smoker
* Previous history of preeclampsia
* Anabolic steroids, cortical steroids, or non-steroidal anti-inflammatory medications, or at the discretion of the investigator.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — transgender women, transgender men, cisgender women, cisgender men on oral and non oral hormone therapy
Study Population: Healthy adult ages 18 - 90 years cisgender (gender identity that aligns with sex at birth) and transgender (gender identity that does not align with sex at birth) adult women and men who are on oral, non-oral or no hormone therapy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
First association in transgender women and cis women | 2025
  to investigate the association between route of administration of exogenous estrogen (transdermal vs. oral) and cardiorenal risk in cisgender (gender identity aligning with sex at birth) and transgender (gender identity not aligning with sex at birth) women.
Second association in transgender men and cis men | 2025
  to investigate the association between exogenous testosterone exposure and cardiorenal risk in cisgender (gender identity aligning with sex at birth) and transgender (gender identity not aligning with sex at birth) men.

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Ahmed, MD, Principal Investigator — Alberta Health services
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No